CLINICAL TRIAL: NCT03253471
Title: A Randomized, Double-blind, Placebo-controlled, First-in-human, 3 Part Study of Orally Administered AL-611 to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics (Part 3) of Single Ascending Doses in Healthy Volunteers (Parts 1-2), and Multiple Ascending Doses in Subjects With Chronic Hepatitis C Virus Infection (Part 3)
Brief Title: A First in Human Study of AL-611 in Healthy Volunteers and Patients With Hepatitis C Virus Infection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic decision to discontinue further development of investigational compounds for the treatment of hepatitis C.
Sponsor: Alios Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL-611-1101
Record Dates: First submitted 2017-08-02; First posted 2017-08-18 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AL-611 (Experimental)
  Interventions: Drug: AL-611
- Placebo to Match AL-611 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AL-611 — AL-611 tablets
  Arms: AL-611
Drug: Placebo — Placebo to Match AL-611
  Arms: Placebo to Match AL-611

SUMMARY:
This randomized, double-blind, placebo-controlled, 3-part study will assess the safety, tolerability, pharmacokinetics (PK), and antiviral activity (Part 3 only) of orally administered AL-611 in healthy volunteers (HV; Parts 1-2) and subjects with CHC (Part 3).

Part 1: HV will receive 1 of 5 single ascending doses (SAD) of AL-611 Part 2: Eight HV from Cohort 3 in Part 1 are planned to receive a second single dose of AL-611 or placebo (as per their randomized assignment in Part 1) in a fed state after a washout period Part 3: Subjects with CHC infection will receive 1 of 3 planned multiple ascending doses (MAD)

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written consent.
* In the investigator's opinion, the subject is able to understand and comply with protocol requirements, instructions, and protocol stated restrictions and is likely to complete the study as planned.
* Except in compensated cirrhosis (cirrhosis cohorts only) and diagnosis of HCV (Part 3 only), subject is in good health as deemed by the investigator, based on the findings of a medical evaluation including medical history, physical examination, laboratory tests, and ECG.
* Male or female, 18-60 years of age for HV and 18-70 years of age for subjects with CHC.
* Body mass index (BMI) 18-30 kg/m2, inclusive, for HV and 18-35 kg/m^2, inclusive, for subjects with CHC. The minimum weight is 50 kg in both populations.
* A female subject is eligible to participate in this study if she is of non-childbearing potential (defined as females with a documented tubal ligation, bilateral oophorectomy, or hysterectomy) or postmenopausal (defined as 12 months of spontaneous amenorrhea and follicle stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal females).
* If male, subject is surgically sterile or practicing specific forms of birth control until 6 months after the end of the study. Male subjects must agree to refrain from sperm donation from start of dosing through 6 months after the completion of study drug administration.
* Subject agrees to refrain from blood donation from screening until 56 days after the last study visit.
* For HV, estimated glomerular filtration rate (eGFR) in the normal range as determined by modification of diet in renal disease (MDRD) formula. For CHC (Part 3) eGFR>60ml/min/1.73m^2 as determined by MDRD (alternative calculations (eg, Cockroft-Gault) may be permissible, if approved by the Sponsor).

Additional inclusion criteria for subjects with CHC infection (Part 3):

* Subjects must have GT1 or GT3 CHC (or GT1-6 for Part 3 optional cohorts) infection identified at screening.
* Documentation of HCV infection for greater than 6 months before randomization as defined by either documented HCV serology demonstrating the presence of anti-HCV antibodies at least 6 months before randomization or documented presence of HCV RNA at least 6 months before randomization.
* Screening HCV RNA viral load ≥50,000 IU/mL (except for subjects with compensated cirrhosis, who may have HCV RNA viral load ≥10^4 IU/mL) using Ampliprep COBAS® Taqman® HCV Test 2.0
* Cirrhotic subjects in Part 3 must have compensated cirrhosis AND meet the Child-Pugh Class A definition AND have a screening Fibroscan with a liver stiffness score>12.5 kPa.

Exclusion Criteria:

1. History or other clinical evidence of significant or unstable cardiac disease (eg, angina, congestive heart failure, myocardial infarction, diastolic dysfunction, significant arrhythmia (eg, long QT syndrome, torsades de pointes), coronary heart disease), moderate to severe valvular disease or poorly controlled hypertension at screening.
2. Family history of prolonged QT syndrome (eg, torsade de pointes) or sudden cardiac death.
3. Clinically significant abnormal screening ECG findings (eg, PR >220 msec, QRS interval >120 msec or corrected QT interval (QTcF) >450 msec for male subjects and >470 msec for female subjects).
4. Participation in either an investigational drug trial or an investigational vaccine trial within 30 days or 5 half lives (whichever is longer) prior to starting study medication.
5. Clinically significant blood loss or elective blood donation of significant volume (ie, >500 mL) within 60 days prior to screening; >1 unit of plasma within 7 days prior to screening.
6. Unwilling to abstain from alcohol for 48 hours prior to the start of dosing through the study completion visit.
7. History of regular alcohol intake >14 units per week of alcohol for females and >21 units per week for males (one unit is defined as 10 g alcohol) within 3 months of randomization
8. The subject has a positive alcohol test at screening or on Day -2.
9. Hypersensitivity to the active substance or to any of the excipients of AL-611
10. Abnormal (using local normal range) heart rate, respiratory rate, temperature or blood pressure (BP) values (evaluated in a semi-recumbent or recumbent position after 5 minutes of rest). One repeat measurement after an additional ~5 minutes of rest is permitted. In addition, a repeat measurement performed on a separate day is also permitted.
11. Clinically significant cardiovascular, respiratory, renal, gastrointestinal, hepatic, hematologic, neurologic, oncologic (except adequately treated basal cell carcinoma and cervical intraepithelial neoplasia [CIN] I or II), autoimmune, or any other medical illness or psychiatric disorder, as determined by the Investigator. CHC with/without compensated cirrhosis acceptable for cohorts enrolling CHC subjects with/without compensated cirrhosis, respectively, but non-HCV related hepatic disease is exclusionary.
12. Positive test for hepatitis A virus (HAV) IgM, hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody. For HV HCV is exclusionary.
13. Evidence of active infection (topical fungal infections which are considered not clinically significant are permitted). CHC is inclusionary for Part 3 only.
14. History of regular use of tobacco (ie, ≥10 cigarettes per day or equivalent for alternative nicotine products (eg, e cigarettes)) within 3 months of randomization.
15. The subject has a positive drug screen during screening or on Day -2. For CHC, prescribed medications with a stable dose for at least 21 days may be considered by the Investigator and Sponsor Medical Monitor; cannabis is permitted.
16. From 14 days (or 5 half-lives, whichever is longer) prior to admission to the Phase 1 Unit until randomization, use of any medications, including prescription, over the counter, and herbal medications, is exclusionary. The only exceptions are acetaminophen, ibuprofen, hormone replacement therapy, and thyroid hormone replacement therapy.
17. Abnormal screening laboratory results that are considered clinically significant by the investigator or as specified in the protocol.

    Additional exclusion criteria for subjects with CHC (Part 3):
18. History of clinical hepatic decompensation, eg, variceal bleeding, spontaneous bacterial peritonitis, ascites, hepatic encephalopathy or active jaundice (within the last year).
19. Except subjects with compensated cirrhosis, a liver biopsy within 2 years that demonstrates cirrhosis (Knodell score >3, Metavir score >3, Ishak score >4) or a screening Fibroscan liver stiffness score >12.5 kPa.
20. Prior treatment for CHC, defined as prior exposure to any approved or investigational drugs intended to treat HCV infection. In subjects with compensated cirrhosis, prior relapse after a complete course of, or premature discontinuation from, interferon-based treatment regimens (±ribavirin) is acceptable, but prior exposure to any direct-acting antivirals (DAAs) is exclusionary.
21. Evidence on screening liver ultrasound of hepatic mass or lesion concerning for malignancy (subjects with cirrhosis only).
22. For CHC subjects without cirrhosis, alpha fetoprotein (AFP) concentrations ≤ upper limit of normal (ULN). If AFP is >ULN, absence of a hepatic mass or lesion must be demonstrated by ultrasound within the screening period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Treatment emergent Adverse events | Up to 21 days
Physical examination findings | Up to 21 days
Incidence and severity of vital sign abnormalities | Up to 21 days
Incidence and severity of 12 lead electrocardiagram abnormalities | Up to 21 days
Incidence and severity of clinical laboratory abnormalities | Up to 21 days

SECONDARY OUTCOMES:
Cmax of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration | Day 1 to Day 8
  PK parameter of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration
C0_h of AL-611 and ALS-022358 (and other metabolites if applicable) following repeat dose administration | Day 1 to Day 21
  PK parameter of AL-611 and ALS-022358 (and other metabolites if applicable) following repeat dose administration
Concentrations in urine of AL-611 and ALS 022358 (and other metabolites if applicable) after a single oral dose | Day 1 to Day 8
  Concentrations in urine of AL-611 and ALS 022358 (and other metabolites if applicable) after a single oral dose in HV in fasted conditions
HCV RNA viral load in subjects with CHC | Screening to Day 21
  HCV RNA viral load (over time, maximum decrease from baseline, and change from baseline over time) in subjects with CHC, defined by GT and host characteristic (eg, presence/absence of compensated cirrhosis)
Sequence analysis of HCV | Day 1 to Day 21
tmax of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration | Day 1 to Day 8
  PK parameter of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration
C24h of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration | Day 1 to Day 8
  PK parameter of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration
Clast of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration | Day 1 to Day 8
  PK parameter of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration
tlast of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration | Day 1 to Day 8
  PK parameter of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration
t1/2 of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration | Day 1 to Day 8
  PK parameter of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration
CL/F of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration | Day 1 to Day 8
  PK parameter of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration
Vz/F of AL-611 following single dose administration | Day 1 to Day 8
  PK parameter of AL-611 following single dose administration
AUC0-inf of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration | Day 1 to Day 8
  PK parameter of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration
AUClast of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration | Day 1 to Day 8
  PK parameter of AL-611 and ALS-022358 (and other metabolites if applicable) following single dose administration
Cmax of AL-611 and ALS-022358 (and other metabolites if applicable) following repeat dose administration | Day 1 to Day 21
  PK parameters of AL-611 and ALS-022358 (and other metabolites if applicable) following repeat dose administration
tmax of AL-611 and ALS-022358 (and other metabolites if applicable) following repeat dose administration | Day 1 to Day 21
  PK parameter of AL-611 and ALS-022358 (and other metabolites if applicable) following repeat dose administration
Cmin of AL-611 and ALS-022358 (and other metabolites if applicable) following repeat dose administration | Day 1 to Day 21
  PK parameters of AL-611 and ALS-022358 (and other metabolites if applicable) following repeat dose administration
t1/2 of AL-611 and ALS-022358 (and other metabolites if applicable) following repeat dose administration | Day 1 to Day 21
  PK parameters of AL-611 and ALS-022358 (and other metabolites if applicable) following repeat dose administration
AUClast of AL-611 and ALS-022358 (and other metabolites if applicable) following repeat dose administration | Day 1 to Day 21
  PK parameters of AL-611 and ALS-022358 (and other metabolites if applicable) following repeat dose administration
AUC0_tau of AL-611 and ALS-022358 (and other metabolites if applicable) following repeat dose administration | Day 1 to Day 21
  PK parameter of AL-611 and ALS-022358 (and other metabolites if applicable) following repeat dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Mina Pastagia, Study Director — Alios Biopharma
Locations (1):
- SGS Life Sciences, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided